CLINICAL TRIAL: NCT03924492
Title: Expanded Access Protocol of ZULRESSO for Adult Patients With Postpartum Depression
Brief Title: Expanded Access Protocol of ZULRESSO™ (Brexanolone) Injection for Adult Patients With Postpartum Depression
Status: Approved for marketing | Type: Expanded Access
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 547-PPD-401
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2019-06

CONDITIONS: Postpartum Depression
Keywords: Expanded Access
MeSH Terms: conditions — Depression, Postpartum | interventions — brexanolone; Injections

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: ZULRESSO (brexanolone) injection — ZULRESSO
  Other Names: Brexanolone; SAGE-547

SUMMARY:
This is an expanded access program intended to provide access to ZULRESSO™ (brexanolone) injection for the treatment of a limited number of eligible women with postpartum depression during the period prior to commercial availability. Requests for access must be made by a healthcare provider for a specific patient based on a determination with patient that the benefits of treatment outweigh the risks and an assessment of eligibility based on program criteria. Sites with eligible patients must apply and meet requirements for participation in the expanded access program.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed an informed consent form prior to any study-specific procedures being performed
2. Subject is an ambulatory female at least 18 years of age
3. Subject agrees to adhere to the study requirements
4. Subject agrees not to be the primary caregiver of any dependents during the infusion
5. Subject must have a negative pregnancy test on Day 1 prior to the start of the ZULRESSO infusion
6. Subject has a current diagnosis of PPD, as assessed by the Investigator

Exclusion Criteria:

1. Subject has end stage renal disease
2. Subject has a known allergy to progesterone or allopregnanolone

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes